CLINICAL TRIAL: NCT06288360
Title: Neoadjuvant Chemotherapy Plus Camrelizumab in PD-L1-negative Locally Advanced Cervical Cancer: a Multicentre, Single-arm, Phase 2 Trial
Brief Title: Neoadjuvant Immunochemotherapy in PD-L1-negative LACC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Southwest Hospital, China (Other); Women's Hospital School Of Medicine Zhejiang University (Other); Anhui Provincial Cancer Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other); Gansu Provincial Maternal and Child Health Care Hospital (Other); Beijing Friendship Hospital (Other); Tianjin Medical University General Hospital (Other); Xiangya Hospital of Central South University (Other); West China Second University Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Zhejiang Cancer Hospital (Other); Shengjing Hospital (Other); Qilu Hospital of Shandong University (Other); Cancer Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Kezhen Li, Prof, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NACI-CERV-002; MA-CervC-II-007 (Other Grant/Funding Number: Jiangsu Hengrui Pharmaceuticals Company Ltd.); [2024](S019) (Other: Ethics Committee of Tongji Medical College, HUST)
Record Dates: First submitted 2024-02-18; First posted 2024-03-01 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-10

CONDITIONS: Cervical Cancer; Locally Advanced Cervical Cancer; PD-L1 Negative; Neoadjuvant Chemoimmunotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — camrelizumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant chemotherapy plus camrelizumab (NACI) (Experimental): Patients first received one cycle of platinum-based doublet priming chemotherapy. After 3 weeks, participants received two cycles of the PD-1 inhibitor camrelizumab combined with chemotherapy every 3 weeks. Patients with stable disease or progressive disease received concurrent chemoradiotherapy, and patients with a complete response or partial response proceeded to radical surgery.
  Interventions: Drug: Camrelizumab; Drug: Paclitaxel-albumin; Drug: Cisplatin; Procedure: radical surgery

INTERVENTIONS:
Drug: Camrelizumab — 200 mg, intravenously, 20-60 min. 2 times, every 21 days
  Other Names: SHR-1210
Drug: Paclitaxel-albumin — 260 mg/m² over 30 min, 3 times, every 21 days
  Other Names: Injectable paclitaxel (albumin bound)
Drug: Cisplatin — 4 h, 75-80 mg/m², 3 times, every 21 days
  Other Names: Cisplatin injection
Procedure: radical surgery — Radical hysterectomy + pelvic lymphadenectomy 士 para-aortic lymphadenectomy

SUMMARY:
This is a multicenter, prospective, single-arm, phase 2 clinical trial designed to evaluate the therapeutic efficacy of the NACI (neoadjuvant chemotherapy plus Camrelizumab) for PD-L1-negative locally advanced cervical cancer.

DETAILED DESCRIPTION:
This multicenter, prospective, single-arm clinical trial is designed to enroll patients with PD-L1-negative, locally advanced cervical cancer. Patients will receive an initial course of priming neoadjuvant chemotherapy, followed by two courses of neoadjuvant immunochemotherapy. The study aims to evaluate the effects of combining neoadjuvant chemotherapy with a PD-1 inhibitor on tumor remission rates, surgical complications, positive margin rates, and patient survival. Additionally, the trial will investigate changes in local immune-related factors and tumor cells during treatment, as well as identify biomarkers that may influence the efficacy of neoadjuvant immunochemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. FIGO 2018 stage IB3, IIA2, or IIB/IIIC1r (tumor size>4cm) cervical cancer and without any treatment (After undergoing gynecological examinations by two associate chief physicians or above, the staging of the patients was determined);
2. Has at least one measurable lesion based on Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1. In principle, the size of the lesion as shown by the magnetic resonance imaging examination is used as the criterion.
3. Histologically confirmed squamous carcinoma, adenocarcinoma (common type) or adenosquamous carcinoma of the cervix;
4. Negative PD-L1 expression on preoperative pathological examination (Combined positive score < 1);
5. 18-70 years of age;
6. Eastern Cooperative Oncology Group score ≤ 1;
7. WBC≥3.5*10^9/L, NEU≥1.5*10^9/L, Platelet≥100×10^9 /L; AST and ALT ≤1.5 times normal upper limit; Total bilirubin ≤1.5 times the upper limit of normal value; serum creatinine and blood urea nitrogen ≤the upper limit of normal value;
8. Well-compliance and willing to keep in touch;
9. Willing to participate in this study, sign the informed consent, and comply with the requirements and limitations outlined in the Informed Consent Form (ICF) and this form.

Exclusion Criteria:

1. Active, known, or suspected autoimmune disease, or a history of an autoimmune disease, except for the following: vitiligo, alopecia areata, Graves's disease, psoriasis, or eczema that has not required systemic therapy within the last 2 years, hypothyroidism that is asymptomatic or requires only stable doses of hormone replacement therapy (due to autoimmune thyroiditis), type 1 diabetes that requires only stable doses of insulin replacement therapy, asthma that subsides completely in childhood and does not require intervention in adulthood, or diseases that do not recur in the absence of external triggers;
2. Prior treatment with immune checkpoint inhibitors, including, but not limited to, other anti-PD-1, anti-PD-L1 antibodies, CTLA-4 antibodies, or antibodies against immune co-stimulators (e.g., antibodies against ICOS, CD40, CD137, GITR, OX40 targets, etc.), or any other therapy targeting a tumor's immune mechanism of action;
3. Known hypersensitivity to any component and/or any excipient of the trial prescribed medication;
4. Immunosuppressive drugs or systemic corticosteroids for immunosuppression (> mg/day of prednisone or other equivalent) within 2 weeks prior to trial dosing; topical, ophthalmic, intra-articular, intranasal, and inhaled corticosteroids are permitted;
5. Received herbs with antitumor effects or drugs with immunomodulatory effects (e.g., thymidine, interferon, interleukin-2) within 2 weeks prior to the trial;
6. Active systemic infection requiring systemic treatment;
7. Serious infection within 4 weeks prior to the first dose, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia;
8. Patients with untreated chronic hepatitis B, or HBV carriers with chronic hepatitis B virus (HBV) DNA greater than 1,000 IU/mL, or patients with active hepatitis C. Inactive HBsAg carriers, patients with hepatitis B who have received treatment and are in stable condition (HBV < 1000 IU/mL), and patients with cured hepatitis C are eligible for enrollment. HCV antibody-positive subjects will be eligible for the study only if they have a negative HCV RNA test;
9. Known active tuberculosis (TB), patients with suspected active TB should undergo chest X-ray and sputum examination in conjunction with clinical signs and symptoms for exclusion;
10. Immunodeficiency or human immunodeficiency virus (HIV antibody positive);
11. Subjects with active inflammatory bowel disease or a history of such disease (e.g., Crohn's disease, ulcerative colitis, or chronic diarrhea). Subjects who are unable to swallow or who have malabsorption syndrome, uncontrolled nausea, vomiting, diarrhea, or other gastrointestinal disorders that severely interfere with drug intake and absorption;
12. Known interstitial lung disease that is symptomatic or may interfere with detection or treatment of immune-associated pneumonia;
13. Treatment with a live or attenuated vaccine administered within 4 weeks prior to the first trial dose, inactivated seasonal influenza virus vaccine is permitted;
14. Have received a prior allogeneic bone marrow transplant or solid organ transplant;
15. History of primary malignant tumor within the last 5 years;
16. Have undergone major surgery (e.g., open abdomen, open chest, organ resection, etc.) and severe trauma within 28 days prior to the first dose of the implantable infusion device is permitted;
17. With a history of gastrointestinal perforation, gastrointestinal fistula, or female genital fistula;
18. Uncontrolled other co-morbidities, symptoms, or medical history, including (i) persons with one of the following cardiovascular diseases or cardiovascular risk factors: myocardial infarction, unstable angina, pulmonary embolism, acute/continuous myocardial ischemia, cerebral vascular accident, transient ischemic attack, or other arterial or venous thrombosis, embolism, or cerebral ischemic event of clinical significance/requiring pharmacologic intervention; and persons who have had, within 6 months, a symptoms of congestive heart failure (New York Heart Association (NYHA) class III and above); (ii) clinically significant bleeding symptoms or a history of significant bleeding characteristics such as gastrointestinal bleeding, gastric ulcer bleeding, or vasculitis within 1 month prior to the first dose; (iii) clinically active hemoptysis, active diverticulitis, abdominal abscesses, and gastrointestinal obstruction; and (iv) uncontrolled pleural effusion, pericardial effusion, or ascites requiring Repeated drainage of ascites; ⑤ Abnormal liver or kidney development or history of surgery;
19. Pregnant or breastfeeding female patients; women of childbearing age who refuse to accept contraceptive measures during neoadjuvant immunotherapy;
20. Concurrent participation in other interventional clinical trials; participation in observational and non-interventional clinical trials is permitted;
21. Any condition that, in the judgment of the investigator, may result in risk in the receipt of the study drug or that would interfere with the evaluation of the safety of the study drug or the interpretation of the study results. Patients who, in the judgment of the Investigator, are unlikely to comply with the study steps, restrictions, and requirements are not permitted to participate in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response | undergoing surgery; up to 2 years.
  Pathologic complete response (pCR) refers to the absence of invasive/in situ cancer in the uterine cervix and/or lymph nodes

SECONDARY OUTCOMES:
Surgical Complications | during and after surgery; an average of 3 years.
  Intraoperative bleeding, vascular injuries, bladder injuries, rectal injuries, and ureteral injuries were measured by the need for suture repair; occlusive nerve injuries were measured by complete severance, and vascular injuries required documentation of the site of injury. Postoperative complications included: cervical stenosis, cervical insufficiency, ureteral/bladder/rectal/vaginal fistula, internal hemorrhage, pelvic infection, lymphocyst, lymphatic fistula, lower extremity edema, lower extremity venous thrombosis, urinary retention, nerve injury, and bowel obstruction.
Objective response rate | measured 3 weeks after the last dose of neoadjuvant treatment and before surgery; up to 2 years.
  the proportion of patients who had either complete response or partial response, assessed by independent central reviewers according to RECIST, version 1.1.
Positive surgical margin rate | undergoing surgery; 2 years
  A positive surgical margin means that cancer cells are present at the edge of the resection specimen.
event-free survival | 7 years
  Event-free survival (EFS) refers to the possibility of experiencing a defined set of events (including progression such as metastasis, death, etc.) following NACI treatment.
overall survival | 7 years
  the time from enrollment to death
adverse event | 7 years
  an event that emerges during treatment having been absent pre-treatment, or worsens relative to the pre-treatment state.
Patient Reported Outcomes | 7 years
  including global quality of life and measures of sexual health

CONTACTS AND LOCATIONS:
Overall Officials: Ding Ma, Study Chair — Tongji Hospital
Locations (12):
- China (12):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Beiing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital (Southwest Hospital), Army Medical University (Third Military Medical University), Chongqing, Chongqing Municipality
  - Gansu Provincial Maternity and Child-care Hospital, Lanzhou, Gansu
  - The Affiliated Tumor Hospital of Guangxi Medical University, Nanning, Guangxi
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Second People's Hospital of Sichuan (Sichuan Cancer Hospital), Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Women's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou Institute of Medicine (HIM), Chinese Academy of Sciences, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No